CLINICAL TRIAL: NCT03687320
Title: Effectiveness and Safety of a Home-Use Low Level Laser Therapy Device as an Adjunct to Standard Treatment Compared to Standard Treatment Alone, for Diabetic Foot Ulcers: A Double Blind, Randomized, Sham-Controlled Clinical Study
Brief Title: Laser Therapy for At-Home Treatment of DIabetic Foot Ulcers
Acronym: LLL&DIAB-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erika Carmel ltd (Other)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TLV-0538-18
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Diabetic Foot Ulcer
Keywords: Photobiomodulation; Low-Level Light Therapy; Low-Level Laser Therapy
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Single center, Prospective, Double Blind, Randomized, Sham-Controlled, Parallel Group, Superiority comparison
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sham control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard and B-Cure Pro (Experimental): Subjects from the Standard and B-Cure Pro group will receive standard care and in addition will self-treat at home daily with the B-Cure device.
  Interventions: Device: B-Cure Pro
- Standard and Sham (Sham Comparator): Subjects from the Standard and sham group will receive standard care and in addition will self-treat at home daily with the sham B-Cure device.
  Interventions: Device: Sham

INTERVENTIONS:
Device: B-Cure Pro — The B-Cure laser Pro is a portal, non-invasive, low level laser therapy device, that emits light in the near infrared (808nm) over an area of 1X4.5 cm2 with power output of 250mW, and energy dose of 5J/min.
  Arms: Standard and B-Cure Pro
Device: Sham — The sham device is externally identical to the B-Cure Pro and emit the same guiding light, but does not emit the therapeutic near infrared rays.
  Arms: Standard and Sham

SUMMARY:
The global prevalence of diabetes is on the rise and with it increase in prevalence of diabetic foot ulcers (DFU). These recalcitrant wounds are difficult to manage and pose a heavy economic burden. Photobiomodulation (low-level laser) is used for acceleration of wound healing.

The current study is designed to evaluate the effectiveness of B-cure laser, a home-use low-level laser device, for acceleration of diabetic foot ulcer healing over standard treatment.

DETAILED DESCRIPTION:
Patients with diabetic foot ulcers will receive standard treatment and in addition will be randomly allocated to receive either active or sham laser device to self-treat at home. The patient's wound will be evaluated every 2 weeks. Adverse events will be documented.

The study hypothesis is that B-Cure laser treatments as an adjunct therapy to standard treatment, applied, at home, by the patient or personal care-giver, can accelerate diabetic foot ulcers healing compared to standard treatment alone.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or Female
4. Age:18-90 years old at the time of Informed Consent (Adult, Senior)
5. Type 1 or type 2 Diabetes Mellitus
6. Presence of a diabetic foot ulcer located in the ankle area or below that has persisted a minimum of 3 months prior to the screening visit
7. Ulcer grade classified as ≤3 according to Wagner grading system or IA according to University of Texas Classification of Diabetic Foot Ulcers.
8. Area of ulcer (after debridement) is at least 4 cm2
9. Arterial perfusion: Patients who demonstrate adequate arterial perfusion defined as either: Ankle/brachial index (ABI) above 0.7 or that have documented confirmation of adequate arterial perfusion
10. Patient and/or caregiver must be able and willing to learn and perform the duties of dressing changes
11. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation

Exclusion Criteria:

1. Pre-existing conditions - evidence of gangrene on any part of affected limb, active Charcot's foot on the study limb; infection at time of screening, deep vein thrombosis (DVT), active malignancy, being on dialysis, anemia (Hb<9 gr/dL)
2. Known allergies to dressing materials, including occlusive dressings and the adhesives on such dressings
3. Scheduled to undergo vascular surgery, angioplasty or thrombolysis at the time of enrollment or history of peripheral vascular repair within 10 weeks of screening
4. History of malignancy on study limb or currently receiving or has received radiation or chemotherapy within 3 months of randomization
5. Taking immunosuppressive medication
6. Received growth factor therapy (e.g., autologous platelet-rich plasma gel, becaplermin, bilayered cell therapy, dermal substitute, extracellular matrix) within two weeks of screening
7. Used oral, or IV antibiotic/antimicrobial agents or medications within 7 days of baseline
8. Has serum albumin level of<3 mg%
9. Presence of ulcers due to other causes not related to diabetes
10. HbA1c > 12% (uncontrolled hyperglycemia)
11. A documented history of alcohol or substance abuse within 6 months of screening
12. Currently enrolled or who have participated, within 30 days of screening, in another investigational device, drug or biological trial that may interfere with study results
13. Pregnant at the time of screening
14. Has any Photobiomodulation (low level laser) device at home

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of complete (100%) wound closure | up to 3 months
  Complete re-epithelialization without drainage

SECONDARY OUTCOMES:
Time to complete (100%) wound closure | up to 3 months
  Time to complete re-epithelialization without drainage

CONTACTS AND LOCATIONS:
Overall Officials: Elchanan Luger, MD, Principal Investigator — Department of Orthopedic Surgery, Sourasky Medical Center, Sackler Faculty of Medicine, Tel Aviv University
Locations (1):
- Department of Orthopedic Surgery, Tel Aviv Sourasky Medical Center, Sackler Faculty of Medicine, Tel Aviv University, Tel Aviv, Israel